CLINICAL TRIAL: NCT06225362
Title: Evaluation and Clinical Outcomes After Routine Cataract Surgery With the Quatera® 700 and the Centurion® Vision System
Brief Title: Quatera 700 vs. Centurion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 23-002
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Quatera 700 (Experimental)
  Interventions: Device: Quatera 700
- Centurion Vision System (Active Comparator)
  Interventions: Device: Centurion

INTERVENTIONS:
Device: Quatera 700 — Phacoemulsification device
  Arms: Quatera 700
Device: Centurion — Phacoemulsification device
  Arms: Centurion Vision System

SUMMARY:
Phacoemulsification is the most common treatment for cataract surgery in the developed countries and over the years it gained importance due to several factors: small incision, surgery performed under topical anesthesia - which reduce injection-related complications - short recovery time, low post operatory induced astigmatism, and low incidence of surgical complications, when compared to the conventional surgeries. The study evaluates 2 different phacoemulsification devices in patients undergoing routine cataract surgery in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing bilateral lens extraction with implantation of a posterior chamber intraocular lens.
* Gender: Males and Females.
* Age: 50 to 80 years old. Solomon KD, DeOliveira A, Sandoval HP 4 CONFIDENTIAL CEP 23-002 Version 1.0/27Jul2023
* Willing and able to provide written informed consent for participation in the study
* Willing and able to comply with scheduled visits and other study procedures.
* Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 1 to 30 days between surgeries
* Subjects requiring an IOL power in the range of +10.0 D to +30.0 D only.
* Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

* Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
* Clinically significant corneal dystrophy.
* Corneal irregularities potentially affecting visual acuity: keratoconus, corneal dystrophy, corneal opacities.
* Endothelial cell count less than 1500 cells/mm2
* History of chronic intraocular inflammation.
* History of retinal detachment.
* Femtosecond arcuates at time of surgery.
* Femtosecond laser assisted cataract surgery in one eye only.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
* Previous intraocular surgery.
* Previous radial keratoromy (RK).
* Previous keratoplasty
* Pupil abnormalities
* Subject who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than YAG capsulotomy, i.e. LASIK)
* Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
* Other ocular procedures at the time of the cataract extraction (i.e., iStent)
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Central corneal thickness | Postoperative day 1
Lens removal time | Intraoperative
  from end of rhexis to complete nucleus removal

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No